CLINICAL TRIAL: NCT05230875
Title: Sexual Dysfunction Among Inflammatory Bowel Disease Adults-Clinical Trial
Acronym: SexIA-CT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2021/16
Record Dates: First submitted 2021-12-02; First posted 2022-02-09 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Inflammatory Bowel Diseases; Crohn Disease; Ulcerative Colitis
Keywords: Inflammatory Bowel Disease; Crohn Disease; Ulcerative colitis; Quality of life; Sexual function
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients participating in the therapeutic education program: Patients participating in an educational program on Inflammatory Bowel Disease (IBD) including a specific discussion on intimacy and sexuality .
  Interventions: Behavioral: self-administered questionnaire
- Patients control (not participating in the therapeutic education program): A control group (at the rate of two controls for one case) will be made up of IBD patients routinely followed in the gastroenterology department.Those patients will not participate in the therapeutic education program.

INTERVENTIONS:
Behavioral: self-administered questionnaire — All patients participating in the therapeutic education program will complete a self-administered questionnaire before participation in educational program.
  A new identical self-questionnaire will be distributed to patients 3 to 6 months after their participation in the therapeutic education program.
  Groups: Patients participating in the therapeutic education program

SUMMARY:
Patients with Inflammatory Bowel Disease (IBD) have higher rates of sexual dysfunction than the general population. We offer an educational program on IBD including a specific discussion on intimacy and sexuality for IBD patients. Our objective is to investigate the benefit of this intervention on sexual function in patients with IBD.

DETAILED DESCRIPTION:
Patients with Inflammatory Bowel Disease (IBD) have higher rates of sexual dysfunction than healthy controls. No interventional study has addressed this matter so far. The aim of our study is to investigative the benefit of a psycho-educational intervention on sexual function in patients with IBD, by comparing patients participating to an educational program including a specific discussion on intimacy and sexuality to patients followed in usual care.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Crohn's disease or Ulcerative Colitis diagnosed according to usual criteria
* Participation to IBD educational program

Exclusion Criteria:

* Unability to read or write French
* Patients without sexual activity for religious reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Crohn's disease or Ulcerative Colitis diagnosed according to usual criteria.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-04-07 (Actual); Primary Completion 2023-09-05 (Estimated); Study Completion 2023-09-05 (Estimated)

PRIMARY OUTCOMES:
Mean scores of sexual function scores using International Index of Erectile Function (IIEF) for men | before participation to educational program
Mean scores of sexual function scores using International Index of Erectile Function (IIEF) for men | from 3 to 6 months after participation to educational program.
Mean scores of sexual function scores using Female Sexual Function Index (FSFI) for women. | before participation to educational program
Mean scores of sexual function scores using Female Sexual Function Index (FSFI) for women. | from 3 to 6 months after participation to educational program.

SECONDARY OUTCOMES:
Mean scores for quality of life (S-IBDQ) | before participation to educational program
Mean scores for quality of life (S-IBDQ) | from 3 to 6 months after participation to educational program.
Mean scores for anxiety and depression (HADS) | before participation to educational program
Mean scores for anxiety and depression (HADS) | from 3 to 6 months after participation to educational program.
Mean scores for fatigue (FSS) | before participation to educational program
Mean scores for fatigue (FSS) | from 3 to 6 months after participation to educational program.
Means score for body image (BIS). | before participation to educational program
Means score for body image (BIS). | from 3 to 6 months after participation to educational program.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Universitaire de Bordeaux, Talence, France

IPD SHARING:
Plan to Share IPD: No